CLINICAL TRIAL: NCT00380848
Title: Effect of Hemodiafiltration on Sleep-Disordered Breathing in Patients With End-Stage Renal Disease
Brief Title: Impact of Different Dialysis on Sleep Apnea in Patients With Renal Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Gambro Renal Products, Inc. (Industry); McGill University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MUHC BMB 05-009
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2006-05

CONDITIONS: Sleep Apnea; End Stage Renal Disease
Keywords: sleep apnea; end stage renal disease; hemodiafiltration
MeSH Terms: conditions — Sleep Apnea Syndromes; Kidney Failure, Chronic | interventions — Hemodiafiltration

INTERVENTIONS:
Procedure: Hemodiafiltration

SUMMARY:
The purpose of this study is to determine whether hemodiafiltration, a new form of hemodialysis can improve sleep apnea in patients with end stage kidney disease.

DETAILED DESCRIPTION:
Sleep apnea or breathing problems during sleep are frequent, occurring in 6% of the general population. However, more than half of all patients on dialysis suffer from breathing problems related to sleep. Sleep apnea is associated with high blood pressure, excessive sleepiness, fatigue, poor memory and concentration as well as depression in those with normal kidneys.

Hemodiafiltration is a new kind of dialysis that is more efficient at clearing toxins that accumulate in kidney failure. It has been used successfully in Europe for over 15 years. However, the effects of hemodiafiltration on sleep apnea in dialysis patients have never been assessed.

We are conducting a clinical trial to examine the effects of hemodiafiltration on sleep apnea in dialysis patients. Fifteen patients with sleep apnea, already on dialysis will be treated with hemodiafiltration 3 times a week, instead of their regular hemodialysis treatment for a period of 3 months. We will repeat sleep studies in these patients before and after the hemodiafiltration period and assess their quality of life.

We hope to decrease the severity of sleep apnea with hemodiafiltration. This could result in better sleep, improved energy level, mood, memory, concentration and blood pressure control in those afflicted by sleep apnea and on dialysis. Our findings would also give us better insight into the cause of sleep apnea in patients with end stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently stable on a thrice weekly hemodialysis regimen for a minimum of 3 months
* Patients with vascular access and no contraindications to anticoagulation
* Presence of sleep-related breathing disorder defined as a mean apnea-hypopnea per hour of recording greater than 10 based on cardiorespiratory monitoring

Exclusion Criteria:

* Patients already on hemodiafiltration therapy
* Patients already on treatment for sleep disordered breathing.
* Patients with significant neuromuscular disease
* Patients with an expected lifespan < 1 year
* Patients unable to complete sleep related quality of life questionnaires and consent forms due to language barriers or dementia
* Patients with known substance abuse
* Patients with a respiratory disturbance index greater than 30 with active cardiovascular disease defined by unstable angina, myocardial infarction within 3 months or an Epworth sleepiness score greater than 15 while actively working in a stress situation (for example bus driver, taxi driver). These patients will be evaluated by a sleep specialist.
* Living further than 30 km from dialysis centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-03; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in apnea hypopnea index after a treatment period of three months of hemodiafiltration; scored on overnight polysomnography

SECONDARY OUTCOMES:
Generic Quality of life
specific quality of life related to sleep apnea
specific quality of life related to Restless leg syndrome
24 hour blood pressure control
Periodic limb movement indices
Validity of a positive screening sleep study
specific quality of life related to sleep
Upper airway neuronal afferent dysfunction
Relationship between cytokine levels and sleep apnea severity
Relationship between dialysis clearance and sleep apnea severity

CONTACTS AND LOCATIONS:
Overall Officials: Kateri A Champagne, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Navdeep Tangri, M.D., Principal Investigator — McGill University; John R Kimoff, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Paul Barre, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Sameena Iqbal, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital - Dialysis Unit, Montreal, Quebec, Canada